CLINICAL TRIAL: NCT00512330
Title: Evaluation of Urine Lipoarabinomannan ELISA In Diagnostics of Childhood Tuberculosis
Brief Title: Lipoarabinomannan (LAM) Enzyme-Linked Immunosorbent Assay (ELISA) in Diagnostics of Childhood Tuberculosis (TB)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Our Lady of Mount Carmel Community Hospital, Kapiri, Malawi (Unknown); Ministry of Health and Population, Malawi (Other Government); Mbeya Medical Research Programme, Mbeya, Tanzania (Unknown); Unterstützerkreis Missionskrankenhaus Kapiri e.V., Munich, Germany (Unknown); Foerderverein AIDS im Kindesalter in Bonn e.V., Bonn, Germany (Unknown); Children's Medical Hospital, University of Bonn, Germany (Other)
Responsible Party: Dr. Norbert Heinrich, Principal Investigator, Department of Tropical Medicine, Ludwig-Maximilan-University, Munich, Germany
Other Study IDs: LAM ELISA in childhood TB
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Tuberculosis
Keywords: childhood; tuberculosis; diagnostic; lipoarabinomannan; ELISA; Tuberculosis in Childhood
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In children, it remains quite difficult even in developed countries, to prove a diagnosis of Tuberculosis (TB). New means for diagnosis of this disease are currently being researched. One candidate test is Lipoarabinomannan ELISA from Urine, which has shown good sensitivity of up to 80% in adults.

Our study aims to evaluate this test in the diagnosis of children with TB.

DETAILED DESCRIPTION:
Among candidate new diagnostics for TB, a test for mycobacterial Lipoarabinomannan (LAM) excretion in urine has shown promising results in one Tanzanian study: The sensitivity for detecting TB culture-positive patients was 80.3%. Of 103 healthy volunteers, only one gave a false positive result (Boehme, 2005).

Until now, there are only data concerning this test for diagnosis of adult disease. For evaluation of routine use in children in countries like Malawi, we are starting a prospective study. Children 0-14 years of age with suspected TB will be investigated using TB culture as the gold standard. In sputum samples, microscopy will be done. Simultaneously, LAM Elisa from the patient´s urine will be done.

ELIGIBILITY:
Inclusion Criteria:

* age 0-14 years
* suspicion of active TB or TB contact

Exclusion Criteria:

* no informed consent

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children up to 14 years of age with suspicion of TB
Enrollment: 250 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Heinrich, MD, Study Chair — University of Bonn; John Chimphamba, Clinical Officer, Principal Investigator — Our Lady of Mount Carmel Hospital, Kapiri; Andreas Mueller, PD Dr med., Study Chair — University of Bonn
Locations (1):
- Our Lady of Mount Carmel Hospital, Kapiri/Mchinji, Mchinji, Malawi